CLINICAL TRIAL: NCT02621073
Title: Does VeraFlo With Prontosan® Decrease Time to Wound and Fracture Healing in Patients With Infected Lower Extremity Fractures With Indwelling Hardware?
Brief Title: VeraFlo With Prontosan® and Wound and Fracture Healing.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was more difficult than expected. It was mutually agreed upon that we would close the study. No results to report.
Sponsor: Brett Crist (Other)
Responsible Party: Sponsor-Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Orthopaedic Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003641
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-05

CONDITIONS: Infection
Keywords: lower extremity; status-post ORIF
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VeraFlo with Prontosan (Active Comparator): V.A.C. VeraFlo™ Therapy, the only NPWT system with an instillation feature which allows solution to dwell in the wound for thorough contact with the wound bed. The solution being instilled is Prontosan: Unlike other antiseptics, the antimicrobial efficacy of Prontosan® is not impaired in human wound fluid, human tissue or by high loads of blood or albumin. Furthermore, Prontosan® blocks the microbial attachment to surfaces and has been shown to effectively remove biofilms in vitro and in vivo (Hubner et al 2010).
  Interventions: Drug: VeraFlo with Prontosan
- V.A.C Ulta System (Active Comparator): The V.A.C.Ulta™ Therapy System is an integrated wound therapy system that provides NPWT (negative pressure wound therapy), without instillation.
  Interventions: Device: V.A.C Ulta System

INTERVENTIONS:
Drug: VeraFlo with Prontosan — VeraFlo device with Prontosan instillation (n=10).
  Arms: VeraFlo with Prontosan
Device: V.A.C Ulta System — V.A.C. Ulta Negative Pressure Wound Therapy System without instillation (n=10).
  Arms: V.A.C Ulta System

SUMMARY:
To answer the question: "Do Prontosan instillations decrease time to wound and fracture healing and decrease bacterial load compared to wound vac treatment without Prontosan?," we will enroll up to 30 subjects (for an anticipated 20 complete data sets) into this trial. The subjects will be split equally into two different groups by randomization. One groups will have wound vac therapy with Prontosan, and one group will have wound vac therapy without Prontosan. Data related to wound and fracture healing and bacterial load will be assessed between the two groups to determine if wound vac therapy with Prontosan speeds up healing time and decreases bacterial load.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are a devastating and relatively common surgical complication, occurring in 2% to 5% of patients undergoing surgery in the United States. SSIs can significantly increase patient morbidity, hospital stay duration, healthcare costs, and patient mortality (Anderson 2011).

Negative Pressure Wound Therapy (NPWT) with Vacuum-Assisted Closure (VAC) is an established adjunctive treatment option for open wounds that offers the ability to promote healing. However, there is limited evidence for its utility with active infections. Wounds that are acutely infected or that contain an adherent biofilm present a challenging problem (Kim et al 2015).

Wound VAC therapy involves cleaning the wound, applying a custom-fit foam to cover the wound, placing a transparent drape over the wound and adjacent skin, and attaching tubing to connect the foam to a VAC suction canister. NPWT is achieved with a pulling force supplied by the VAC suction canister. Typically, suction will remain at a constant pressure until the dressing is removed. Continuous VAC therapy was recently reported to be more effective than standard moist wound care in surgical site infection after ankle surgery (Zhou et al. 2015).

VAC therapy with instillations is a novel treatment option that provides the combination of negative pressure with intermittent instillation of a solution. Polihexanide (Prontosan®) is a modern antiseptic that combines a broad antimicrobial spectrum with low toxicity, high tissue compatibility, no reported adsorption and good applicability as solution, gel, ointment, foam and in wound dressing. Unlike other antiseptics, the antimicrobial efficacy of Prontosan® is not impaired in human wound fluid, human tissue or by high loads of blood or albumin. Furthermore, Prontosan® blocks the microbial attachment to surfaces and has been shown to effectively remove biofilms in vitro and in vivo (Hubner et al 2010).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Patients who will be undergoing surgical management (including the use of NPWT therapy) of an infected lower extremity status-post open reduction and internal fixation (ORIF)

Exclusion Criteria:

* Pregnant females
* Incarcerated patients and those not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Crist, MD, Principal Investigator — University of Missouri, Missouri Orthopaedic Institute
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VeraFlo With Prontosan: VeraFlo with Prontosan: VeraFlo device with Prontosan instillation.
- V.A.C Ulta System: V.A.C Ulta System: V.A.C. Ulta Negative Pressure Wound Therapy System without instillation
Period: Overall Study
Arm/Group | VeraFlo With Prontosan | V.A.C Ulta System
Started | 4 | 3
Completed | 1 | 0
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VeraFlo With Prontosan | V.A.C Ulta System | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 51.25 [37 to 64] | 59.3 [55 to 66] | 54.7 [37 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Full Range); unit: kg/m^2] | 35.8 [24 to 57] | 28.3 [24 to 33] | 32.6 [24 to 57]

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Load
Description: Semiquantitative wound culture(s) done at each debridement procedure, (up to 3). Organism quantities are listed as scant, moderate, or heavy. Report includes identification of organism, and susceptibility. Wound cultures will be analyzed and reported by the University of Missouri Hospital Laboratory.
Time Frame: approximately 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VeraFlo With Prontosan | V.A.C Ulta System
Number analyzed (Participants) | 4 | 3
Participants
  No Bacterial Growth | 1 | 0
  Scant Bacterial Growth | 1 | 1
  Moderate Bacterial Growth | 1 | 1
  Heavy Bacterial Growth | 1 | 1

2. Secondary Outcome: Number of Operative Debridements Until Wound Healed
Time Frame: 12 months
Measure: Mean (Full Range); unit: Operations
Arm/Group | VeraFlo With Prontosan | V.A.C Ulta System
Number analyzed (Participants) | 4 | 3
Operations | 2.3 [2 to 3] | 2.3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | VeraFlo With Prontosan | V.A.C Ulta System
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeraFlo With Prontosan (N=4) | V.A.C Ulta System (N=3)
Below Knee Amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deep Surgical Site Infection (Infections and infestations) | 3 (3) | 0 (0)
Syndesmosis Rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-12-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT02621073/Prot_000.pdf